CLINICAL TRIAL: NCT01826500
Title: VARITI-5 : Study of Variations of Serum ITIH5 in Women During the Genital Life and in Pathological Situations.
Acronym: VARITI-5
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LOC/12-16 - VARITI-5; 2012-A01470-43 (Other: ID RCB); 121347B-22 (Other: ANSM); 12/45-878 (Other: CPP Rennes Ouest V)
Record Dates: First submitted 2013-03-25; First posted 2013-04-08 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: IVF; Endometriosis
Keywords: embryo transfer; IVF cycle; endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients having any of the following criteria:
  * Patients with embryo transfer fresh or frozen
  * Patients from an IVF cycle,
  * Patients supported surgically for endometriosis
  Interventions: Other: blood test
- Controls: Controls
  Interventions: Other: blood test

INTERVENTIONS:
Other: blood test — blood test

SUMMARY:
The five proteins of the ITI (Inter-α-trypsin inhibitor) family, are essential components of the extracellular matrix, the dynamics of which they participate in the processes of cellular differentiation and proliferation. I. The ITIH1, ITIH2, ITIH3 and ITIH4 genes seem to be overwhelmingly expressed in the liver, this organ secreting then the corresponding proteins in the general circulation. The only data on ITIH5 indicate that this gene is poorly expressed in the liver and that the major source of its expression is the placenta. In the context of genetic studies on the syndrome of Mayer-Rokitansky-Küster-Hauser (congenital aplasia of the uterus and vagina), the investigators have shown the involvement of ITIH5 and implemented validation experiments of this gene in mice. The investigators have shown that the production of ITIH5 by the uterus varies greatly depending on the physiological state of this organ, especially during pregnancy and the estrous cycle. The investigators also found that most of the production ITIH5 was located in the uterus. Therefore, the serum dosage of ITIH5 could be used clinically as a new biological marker specific to the uterus. This non-invasive biological marker could thus assist in the diagnosis and the understanding of uterine pathologies. ITIH5 rate being correlated to endometrial proliferation, its dosage could be an early and non-invasive marker of endometriosis. The peak of production of ITIH5 by the uterus at the time of embryo implantation window indicates that the assay could provide a better assessment of endometrial receptivity to embryo. It then could be a hand tool of diagnosis in some cases of early repeated miscarriages, and secondly, a prognostic tool for embryo implantation in the context of in vitro fertilization.

The investigators conducted an initial feasibility study on the serum dosage of ITIH5, which was approved by the ethics committee of the University Hospital of Rennes. This first step has been validated. Now, the project is to perform a quantitative analysis of ITIH5 and to correlate clinical and biological data of relevant pathological and physiological situations. This project was the subject of a national and international patents of which the University Hospital of Rennes is promoter.

DETAILED DESCRIPTION:
Pilot study, prospective, single-center, biomedical

ELIGIBILITY:
Inclusion Criteria:

For patients

* Patients having any of the following criteria:
* Patients with embryo transfer fresh or frozen
* Patients from an IVF cycle,
* Patients supported surgically for endometriosis Age between 18 and 45 years, Subjects affiliated to the social security Having given free and informed consent in writing.

For donors

* Aged between 18 and 45 years,
* Subjects affiliated to the social security
* Having given free and informed consent in writing.

Exclusion Criteria:

For patients

For all patients:

* Subjects under 18 years (minors)
* The majors protected (judicial protection, guardianship and curatorship) and persons deprived of their liberty,
* Patients with cancer of gynaecological origin or not,
* Patients with acute or chronic liver disease.

For patients with embryo transfer:

- Patients with endometriosis.

For patients with endometriosis:

- Hormonal treatment for endometriosis in progress.

For donors

For all donors:

* Subjects under 18 years (minors)
* The majors protected (judicial protection, guardianship and curatorship) and persons deprived of their liberty,
* Patients with cancer of gynaecological origin or not,
* Patients with acute or chronic liver disease.

For female subjects:

* Taking hormonal contraception whatever the pharmaceutical or any other œstro-progestative treatment,
* Past or present support in Medically Assisted Reproduction,
* Subjects with an ongoing pregnancy,
* Subjects with endometriosis
* Menopausal subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients with embryo transfer fresh or frozen
  * Patients from an IVF cycle,
  * Patients supported surgically for endometriosis or
  * donors
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2013-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Serum levels of the protein ITIH5 | Day 1
  To establish the normal serum levels of the protein ITIH5 during the life female genital

SECONDARY OUTCOMES:
Serum levels of the protein ITIH5 of healthy volunteers. | Day 1
  Serum levels of the protein ITIH5 of healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Karine Morcel, MD, Principal Investigator — Rennes University Hospital
Locations (2):
- France (2):
  - EFS de Bretagne, Rennes, Britanny
  - Rennes University Hospital - Hôpital Sud, Rennes, Britanny